CLINICAL TRIAL: NCT01763593
Title: A Prospective, Open Label, Observational Study To Evaluate The Safety And Surgical Performance Of Surgical Blade (Aurosleek) In Cataract Patients
Brief Title: Safety and Surgical Performance Study of Aurosleek Surgical Blades
Acronym: Aurosleek
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aurolab (Other)
Responsible Party: Sponsor
Other Study IDs: AUROSLEEK/CIP/001/2012
Record Dates: First submitted 2012-12-25; First posted 2013-01-09 (Estimated); Last update posted 2013-04-30 (Estimated); Status verified 2013-04

CONDITIONS: Cataract
Keywords: Patients having cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Aurosleek blades: Patients having cataract will undergo surgery by using Aurosleek blades

SUMMARY:
To evaluate the safety and surgical effectiveness of surgical blades (Aurosleek) made by Aurolab.

DETAILED DESCRIPTION:
Cataract till today remains the most common yet treatable cause of blindness accounting for more than 50% of blindness and visual impairment in the developing world. One of the most important features of a blade for cataract surgery is its predictable and repeatable behavior. The surgeon repeatedly and reliably needs to create similar tunnels of the proper length. Aurolab is producing surgical blades (Aurosleek) intended for making incision in cataract surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Senile cataract
* Willing to give written informed consent
* Ability to follow study instructions and likely to complete required visits.

Exclusion Criteria:

* Intraoperative complication including Posterior Capsular Rent and Zonular dialysis
* Traumatic cataract
* Uveitis and Complicated cataract
* One eyed patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cataract surgery would be included in this observational study
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-05 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Physioclinical Characters | 30 days
  Assessment of physio-clinical characteristics of surgical blade such as handling of the blade, sharpness and smoothness of blade.
  Handling of the surgical blade will be assessed in grades of difficult to handle,easy to handle and very easy to handle intraoperatively. Sharpness and smoothness of the blade will be rated as poor or optimum while performing cataract surgery.

SECONDARY OUTCOMES:
Post operative complications | 30 days
  The frequency and occurrence of post operative complications such as rhexis tear, posterior capsular rupture, severe corneal edema, severe iritis and anterior vitrectomy.
  Post operative complications occurrence due to surgical blade will be observed and graded as none or mild or moderate or severe at surgery and post operative 30 days.

CONTACTS AND LOCATIONS:
Overall Officials: Neeraj Kumar Agrawal, MS, Principal Investigator — Medical Officer
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India